CLINICAL TRIAL: NCT06922591
Title: A Phase 1/2, Multicenter, Open-Label Study to Evaluate Safety, Tolerability & Antitumor Activity of TNG462 in Combination With Other Agents in Patients With Pancreatic Cancer With MTAP Loss and Pancreatic or Non-Small Cell Lung Cancer With MTAP Loss & RAS Mutation
Brief Title: Study to Evaluate the Safety, Tolerability & Efficacy of TNG462 in Combination in PDAC & NSCLC Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tango Therapeutics, Inc. (Industry)
Collaborators: Revolution Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TNG462-C102
Record Dates: First submitted 2025-03-28; First posted 2025-04-10 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: PDAC; PDAC - Pancreatic Ductal Adenocarcinoma; NSCLC; RAS Mutation; MTAP Deletion; Lung Cancer; Pancreatic Cancer Metastatic; Thoracic Cancer
Keywords: PRMT5 inhibitor; RAS G12D; Multi RAS; RMC-9805; RMC-6236; Thoracic; Targeted therapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose escalation of TNG462 + RMC-9805, TNG462 + RMC-6236, TNG462 + mFOLFIRINOX and TNG462 + gemcitabine/nab-paclitaxel, followed by expansion of each combination in MTAP loss and RAS mutant PDAC and NSCLC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Escalation 1A (Experimental): Escalating oral doses of TNG462 in combination with oral RMC-6236
  Interventions: Drug: TNG462; Drug: RMC-6236
- Dose escalation 1B (Experimental): Escalating oral doses of TNG462 in combination with oral RMC-9805
  Interventions: Drug: TNG462; Drug: RMC-9805
- Dose Expansion 2A (Experimental): Expansion arm at the RDE(s) of oral TNG462 in combination with oral RMC-6236
  Interventions: Drug: TNG462; Drug: RMC-6236
- Dose Expansion 2B (Experimental): Expansion arm at the RDE(s) of oral TNG462 in combination with oralRMC-9805
  Interventions: Drug: TNG462; Drug: RMC-9805
- Experimental: Dose Escalation 1C (Experimental): Escalating doses of TNG462 in combination with mFOLFIRINOX
  Interventions: Drug: TNG462; Drug: mFOLFIRINOX
- Experimental: Dose Escalation 1D (Experimental): Escalating doses of TNG462 in combination with gemcitabine/nab-paclitaxel
  Interventions: Drug: TNG462; Drug: gemcitabine/nab-paclitaxel
- Experimental: Dose Expansion 2C (Experimental): Expansion arm at the RDE(s) of TNG462 in combination with mFOLFIRINOX
  Interventions: Drug: TNG462; Drug: mFOLFIRINOX
- Experimental: Dose Expansion 2D (Experimental): Expansion arm at the RDE(s) of TNG462 in combination with gemcitabine/nab-paclitaxel
  Interventions: Drug: TNG462; Drug: gemcitabine/nab-paclitaxel

INTERVENTIONS:
Drug: TNG462 — MTA cooperative PRMT5 inhibitor
Drug: RMC-9805 — RAS(ON) G12D selective covalent inhibitor
  Arms: Dose Expansion 2B; Dose escalation 1B
Drug: RMC-6236 — RAS(ON) multi-selective inhibitor
  Arms: Dose Escalation 1A; Dose Expansion 2A
Drug: mFOLFIRINOX — Chemotherapy
  Arms: Experimental: Dose Escalation 1C; Experimental: Dose Expansion 2C
Drug: gemcitabine/nab-paclitaxel — Chemotherapy
  Arms: Experimental: Dose Escalation 1D; Experimental: Dose Expansion 2D

SUMMARY:
TNG462-C102 is a Phase 1/2, open-label, multicenter study designed to determine the safety, tolerability, PK, PD, and preliminary antineoplastic activity of oral TNG462 in combination with RMC-6236, RMC-9805, mFOLFIRINOX or gemcitabine/nab-paclitaxel. The study comprises a dose escalation phase and a dose expansion phase.

DETAILED DESCRIPTION:
TNG462-C102 is a Phase 1/2, open-label, multicenter study designed to determine the safety, tolerability, PK, PD, and preliminary antineoplastic activity of oral TNG462 in combination with RMC-6236, RMC-9805, mFOLFIRINOX or gemcitabine/nab-paclitaxel.

For the RAS inhibitor arms, the study will be conducted in patients with MTAP loss and RAS mutant metastatic pancreatic adenocarcinoma (PDAC) or locally advanced or metastatic non-small cell lung cancer (NSCLC). For the chemotherapy specific arms, the study will be conducted in patients with MTAP loss locally advanced or metastatic PDAC. The entire study (all arms) will be conducted in 2 parts: Phase 1 (dose escalation) and Phase 2 (dose expansion).

Individual Arms in the dose expansion phase may open once the MTD and/or RD(s) has been determined for the corresponding combination in the dose escalation phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Is ≥18 years of age at the time of signature of the main study ICF.
2. Has an ECOG PS of 0 or 1.
3. Has a tumor with loss of MTAP protein or bi-allelic deletion of the MTAP gene
4. Arms A and B only: Has a tumor with a RAS mutation
5. Pathologically documented metastatic PDAC or locally advanced, recurrent or metastatic NSCLC
6. Has received prior standard therapy
7. Arms A and B only: Must not have received prior RAS-targeted therapy
8. Has evidence of measurable disease based on RECIST v1.1.
9. Adequate organ function
10. Must be able to swallow tablets.
11. Negative pregnancy test at screening
12. Written informed consent must be obtained according to local guidelines

Exclusion Criteria:

1. Has received prior treatment with a PRMT5 inhibitor, or MAT2A inhibitor
2. Arms A and B only: Prior enrollment in any phase 3 clinical trial of RMC-6236 or RMC-9805
3. Known allergy, hypersensitivity or intolerance to TNG462 (all arms), RMC-6236 Arm A), RMC-9805 (Arm B), mFOLFIRINOX (Arm C), gemcitabine/nab-paclitaxel (Arm D) or their excipients
4. Has uncontrolled intercurrent illness that will limit compliance with the study requirements.
5. Has an active infection requiring systemic therapy.
6. Is currently participating in or has planned concurrent participation in a study of another investigational agent or device.
7. Has impairment of GI function or disease that may significantly alter the absorption of the oral medications
8. Has known or suspected active or untreated CNS metastases associated with progressive neurological symptoms
9. Has current active liver disease from any cause
10. Is known to be HIV positive, unless all the following criteria are met:

    1. CD4+ count ≥300/µL.
    2. Undetectable viral load.
    3. Receiving highly active antiretroviral therapy
11. Has clinically relevant cardiovascular disease
12. History of or presence of active interstitial lung disease
13. Is a female patient who is pregnant or lactating
14. Is unwilling or unable to comply with the scheduled visits, study treatment administration plan, laboratory tests or other study procedures and study restrictions.
15. Has a prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the investigator's opinion may affect the safety of the patient or impair the ability to assess study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Maximum Tolerated Dose | 21 days
  To determine the MTD and RD(s) of TNG462 in combination with RMC-6236 or RMC-9805
Phase 1: Maximum Tolerated Dose | 28 days
  To determine the MTD and RD(s) of TNG462 in combination with mFOLFIRINOX or gemcitabine/nab-paclitaxel
Phase 2: Combination Anti-neoplastic Activity | 12 weeks
  To assess preliminary evidence of antineoplastic activity of TNG462 in combination with RMC-6236, RMC-9805, mFOLFIRINOX or gemcitabine/nab-paclitaxel using RECIST 1.1

SECONDARY OUTCOMES:
Phase 1: Combination Anti-neoplastic Activity | 12 weeks
  To assess preliminary evidence of antineoplastic activity of TNG462 in combination with RMC-6236, RMC-9805, mFOLFIRINOX, or gemcitabine/nab paclitaxel using RECIST 1.1
Phase 1 and 2: Tmax of TNG462 and in Combination | 21 days
  To characterize the Tmax of TNG462 in combination with RMC-6236 or RMC-9805
Phase 1 and 2: Tmax of TNG462 and in Combination | 28 days
  To characterize the Tmax of TNG462 in combination with mFOLFIRINOX, or gemcitabine/nab-paclitaxel
Phase 1 and 2: Cmax of TNG462 and in Combination | 21 days
  To characterize the Cmax of TNG462 in combination with RMC-6236 or RMC-9805
Phase 1 and 2: Cmax of TNG462 and in Combination | 28 days
  To characterize the Cmax of TNG462 in combination with mFOLFIRINOX, or gemcitabine/nab-paclitaxel
Phase 1 and 2: AUC of TNG462 and in Combination | 21 days
  To characterize the AUC of TNG462 and in combination with RMC-6236 or RMC-9805
Phase 1 and 2: AUC of TNG462 and in Combination | 28 days
  To characterize the AUC of TNG462 in combination with mFOLFIRINOX, or gemcitabine/nab-paclitaxel
Phase 1 and 2 Adverse Event Profile | 21 days
  To determine the safety and tolerability of TNG462 in combination with RMC-6236 or RMC-9805
Phase 1 and 2 Adverse Event Profile | 28 days
  To determine the safety and tolerability of TNG462 in combination with mFOLFIRINOX or gemcitabine nab-paclitaxel

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Pimpkin, MD, PhD, Study Director — Tango Therapeutics, Inc.
Locations (12):
- United States (12):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Sarah Cannon Research Institute Denver, Denver, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Indiana, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Dallas, Irving, Texas
  - NEXT Oncology, Fairfax, Virginia